CLINICAL TRIAL: NCT00418236
Title: Evaluation of Changes in Mammographic Breast Density Associated With Bazedoxifene, Raloxifene, and Placebo in Postmenopausal Women: An Ancillary Study of Protocol 3068A1-301-WW
Brief Title: Effect of Bazedoxifene, Raloxifene, and Placebo on Breast Density
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 3068A1-400
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2007-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
It has been shown that women who have dense breasts have an increased risk of breast cancer compared with women whose breasts are less dense. However, while breast density may be a risk factor, the etiology of the relationship between breast cancer and breast density is not understood. Furthermore, it is well recognized that breast cancer can still develop in women whose breasts are not dense.

At menopause, the amount of breast glandular tissue and stroma naturally decreases due to a lack of hormonal stimulation. This is characterized as a decrease in the mammographic density. Although certain medications, including hormone therapy (HT) and dopamine antagonists can increase breast density, these effects are reversible upon discontinuation of the specific agent. Other medications such as the selective estrogen receptor modulators (SERM), raloxifene (RAL) and tamoxifen, have been shown to not affect breast density and allow the normal age-related changes to occur. The effects of bazedoxifene (BZA), a new SERM, on breast density are not known. The purpose of this study is to examine the effect of BZA on breast density changes over 24 months in postmenopausal women. The results may be useful for clinicians to understand the effect of BZA on breast density and its mammographic effects.

This is an observational, multicenter, double-blind, randomized, placebo- and active comparator-controlled study. It is also an ancillary that will use women who are already participants in a phase 3 trial for fracture reduction (protocol 3068A1-301-WW; primary study). In the primary study, subjects received BZA 20 mg, BZA 40 mg, RAL 60 mg, or placebo. This ancillary study will request a subset of participants to use their mammograms taken in this study. Their mammogram will be digitized by a central imaging center. A single radiologist will perform the quantifications of breast density from the digitized mammograms.

ELIGIBILITY:
1. Each subject must have participated or is currently participating in study 3068A1 301, and must satisfy all of the following criteria
2. Has completed 24 months of treatment.
3. Had a mammogram at the baseline visit and at the month 24 visit, and both are original films that are technically acceptable for reading.
4. Was less than or equal to 62 years of age at the time of study randomization in the primary study.
5. Was at least 80% compliant with test article administration.
6. Did not take any medications 6 months prior to screening in the primary study or during the first 24 months of the study that could cause a change in breast density.
7. Was enrolled at a site that has at least 4 subjects meeting all of the above inclusion criteria.
8. Was enrolled at a clinical site that is still participating in the primary study.

Ages: 18 Years to 63 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400
Dates: Start 2006-10; Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Bulgaria, WVPIMED@wyeth.com; Trial Manager, Principal Investigator — For Croatia, WPBUMED@wyeth.com; Trial Manager, Principal Investigator — For Denmark, medinfonord@wyeth.com; Trial Manager, Principal Investigator — For Estonia, WVPMED@wyeth.com; Trial Manager, Principal Investigator — For Netherlands, trials-NL@wyeth.com; Trial Manager, Principal Investigator — For Poland, WPWZMED@wyeth.com; Trial Manager, Principal Investigator — For Romania, WVPIMED@wyeth.com; Trial Manager, Principal Investigator — For South Africa, ZAFinfo@wyeth.com; Trial Manager, Principal Investigator — For Canada, clintrialparticipation@wyeth.com; Trial Manager, Principal Investigator — For Mexico, gomezzlj@wyeth.com; Trial Manager, Principal Investigator — For Argentina, Scheima@wyeth.com; Trial Manager, Principal Investigator — For Chile, scheima@wyeth.com; Trial Manager, Principal Investigator — For Brazil, xavierl@wyeth.com
Locations (36):
- United States (10):
  - San Diego, California
  - Upland, California
  - Meridian, Idaho
  - Brooklyn Center, Minnesota
  - Billings, Montana
  - Bozeman, Montana
  - Bismarck, North Dakota
  - Fargo, North Dakota
  - Jamestown, North Dakota
  - Watertown, South Dakota
- Buenos Aires, Argentina
- Brazil (3):
  - Sorocaba, São Paulo
  - Goiânia
  - Mato Grosso
- Sofia, Bulgaria
- Canada (4):
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Québec, Quebec
  - Sherbrooke, Quebec
- Santiago, Chile
- Croatia (2):
  - Zadar
  - Zagreb
- Vejle, Denmark
- Estonia (2):
  - Tallinn
  - Tartu
- Agarismo, Mexico
- Amsterdam, Netherlands
- Poland (2):
  - Krakow
  - Warsaw
- Romania (3):
  - Bucharest
  - Cluj-Napoca
  - Iasi, Jud. Iasi
- South Africa (4):
  - Johannesburg
  - Parow
  - Pretoria
  - Somerset West